CLINICAL TRIAL: NCT04501744
Title: A Phase 1, Multicenter, Open-label, Dose-escalation Study to Evaluate the Safety, Tolerability and PK/PD of Recombinant Anti-EpCAM and Anti-CD3 Human-Mouse Chimeric Bispecific Antibody Via Intraperitoneal Infusion in Malignant Ascites
Brief Title: A Study of M701 (EpCAM and CD3) in Malignant Ascites
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wuhan YZY Biopharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M70101
Record Dates: First submitted 2020-07-17; First posted 2020-08-06 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Malignant Ascites; Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- M701 (Experimental): Patients will undergo a 2-week screening period and a 4-week core treatment period, and eligible patients who complete the core treatment period will receive a cycle of extended treatment (once weekly for 4 weeks) until disease progression or toxicity intolerance.
  Interventions: Drug: Cohort 1 of M701; Drug: Cohort 2 of M701; Drug: Cohort 3 of M701; Drug: Cohort 4 of M701; Drug: Cohort 5 of M701; Drug: Cohort 6 of M701; Drug: Cohort 7 of M701

INTERVENTIONS:
Drug: Cohort 1 of M701 — Patients in Cohort 1 will receive 4 escalating doses (2, 5, 10 and 25 μg) of M701 on Days 1, 8, 15 and 22. The maintenance dose during extended treatment period is 25 μg.
Drug: Cohort 2 of M701 — Patients in Cohort 2 will receive a starting dose on Day 1 and three infusions at a higher maintenance dose level on Days 8, 15 and 22. The starting dose is 25 μg, and the maintenance dose during core treatment period and extended treatment period is 50 μg.
Drug: Cohort 3 of M701 — Patients in Cohort 3 will receive a starting dose on Day 1 and three infusions at a higher maintenance dose level on Days 8, 15 and 22. The starting dose is 50 μg, and the maintenance dose during core treatment period and extended treatment period is 100 μg.
Drug: Cohort 4 of M701 — Patients in Cohort 4 will receive a starting dose on Day 1 and three infusions at a higher maintenance dose level on Days 8, 15 and 22. The starting dose is 100 μg, and the maintenance dose during core treatment period and extended treatment period is 200 μg.
Drug: Cohort 5 of M701 — Patients in Cohort 5 will receive a starting dose on Day 1 and three infusions at a higher maintenance dose level on Days 8, 15 and 22. The starting dose is 150 μg, and the maintenance dose during core treatment period and extended treatment period is 300 μg.
Drug: Cohort 6 of M701 — Patients in Cohort 6 will receive a starting dose on Day 1 and three infusions at a higher maintenance dose level on Days 8, 15 and 22. The starting dose is 200 μg, and the maintenance dose during core treatment period and extended treatment period is 400 μg.
Drug: Cohort 7 of M701 — Patients in Cohort 7 will receive a starting doseon Day 1 and three infusions at a higher maintenance dose level on Days 8, 15 and 22. The starting dose is 250 μg, and the maintenance dose during core treatment period and extended treatment period is 500 μg.

SUMMARY:
This study is to investigate the safety, tolerability, PK, PD and immunogenicity of multiple ascending doses of M701 administered intraperitoneally to patients with malignant ascites caused by advanced solid tumors.

DETAILED DESCRIPTION:
To evaluate the safety and tolerability of multiple ascending doses of M701 administered intraperitoneally in patients with malignant ascites.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females, aged > 18 years;
2. Histologically- or cytologically-confirmed advanced solid tumors;
3. Patients who require therapeutic paracentesis, defined as at least 1 therapeutic paracentesis (e.g., to relieve abdominal pressure and discomfort) during 4 weeks prior to the baseline paracentesis;
4. Patients who have failed to standard treatment, or who have no standard treatment available that may confer clinical benefit;
5. EpCAM+ tumor cells in ascites fluid;
6. Patients who have received anti-tumor therapy including chemotherapy, hormone therapy, radiotherapy (except local radiotherapy for pain relief) ≥ 2 weeks or received immunotherapy, biological agents ≥ 3 weeks prior to the first dose of study drug;
7. Patients who have recovered from any toxic reaction to previous medications (Grade 0 or 1 based on NCI-CTCAE v5.0);
8. Patients with an ECOG Performance Status score (PS) 0-3;
9. Patients with a life expectancy > 8 weeks;
10. Organ function levels must meet the following requirements:

    Bone marrow: absolute neutrophil count (ANC) ≥ 1.5 ×10^9/L, platelet count ≥ 80 ×10^9/L, hemoglobin ≥ 9.0 g/dL (without blood transfusion within14 days of the first dose of study drug); Liver: bilirubin ≤ 1.5 x upper limit of normal (ULN), aspartate aminotransferase (AST) and alanine transaminase (ALT) ≤ 3 x ULN ( ≤ 5 x ULN in case of liver metastases); Kidney: serum creatinine ≤1.5 x ULN and estimated glomerular filtration rate (eGFR) ≥ 50 ml/min;
11. Patients must understand and voluntarily sign the informed consent form.

Exclusion Criteria:

1. Known to have a history of allergy to the active ingredients of M701; or with a definite history of drug allergy or specific allergy (asthma, rubella, eczema dermatitis);
2. Known or suspected hypersensitivity to M701 or similar antibodies;
3. Extensive liver metastases (> 70% organ volume comprises malignancy);
4. Uncontrolled active infection (CTCAE ≥ Grade 2);
5. Serious diarrhea (CTCAE ≥ Grade 2);
6. Serious dyspnea requiring oxygen therapy;
7. History of auto-immune diseases (e.g. inflammatory bowel disease, idiopathic thrombocytopenic purpura, lupus erythematosus, autoimmune hemolytic anemia, scleroderma, serious psoriasis, rheumatoid arthritis);
8. History of acute or chronic pancreatitis;
9. Other serious diseases that may prevent patients participation in this trial (such as uncontrolled diabetes mellitus, severe gastrointestinal disorders);
10. Cardiac insufficiency, NYHA class III or IV;
11. Intestinal obstruction that occurred within 30 days prior to the first dose of study drug;
12. Non-drainable ascites;
13. Confirmed portal vein obstruction;
14. History of immunodeficiency, including positive HIV test;
15. Active hepatitis B virus infection or hepatitis C virus infection, positive syphilis antibody test and positive HIV antibody test;
16. Pregnant or breastfeeding woman;
17. Plan to conceive within six months;
18. Previous confirmed history of neurological or mental disorders, including epilepsy and dementia;
19. Have received a clinical study active drug treatment within 1 month prior to the first dose of study drug;
20. Those that are deemed ineligible for this clinical trial by study personnel.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2018-09-30 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
MTD | From the time of the first dose (Day 1) until the forth dosing (Day 28)
  Number of DLTs (dose limiting toxicities) during the first 28 days after the first administrations of study drug in each cohort.
Incidence of AEs | From the start of administration to the end of the study or 28 days after the administration is stopped (up to 6 months and 28 days)
  Incidence and severity of AEs, including but not limited to vital signs, physical examination, laboratory tests. All AEs will be classified as Grades 1 through 5 as defined by NCI CTCAE v5.0.

SECONDARY OUTCOMES:
Area under the curve (AUC) of M701 | From the time of first dosing (Day 1) until disease progression or toxicity intolerance (up to 6 months).
  The endpoints for assessment of PK of M701 include serum concentrations of M701 at different timepoints after M701 administration.
Maximum observed concentration (Cmax) of M701 | From the time of first dosing (Day 1) until disease progression or toxicity intolerance (up to 6 months).
  The endpoints for assessment of PK of M701 include serum concentrations of M701 at different timepoints after M701 administration.
Minimum observed concentration (Cmin) of M701 | From the time of first dosing (Day 1) until disease progression or toxicity intolerance (up to 6 months).
  The endpoints for assessment of PK of M701 include serum concentrations of M701 at different timepoints after M701 administration.
The antibody titer of the neutralizing antibody | From the time of first dosing (Day 1) until disease progression or toxicity intolerance (up to 6 months).
  The immunogenicity of M701 will be collected by testing the antibody titer of the neutralizing antibody.
Number of subjects who develop detectable anti-drug antibodies (ADAs) | From the time of first dosing (Day 1) until disease progression or toxicity intolerance (up to 6 months).
  The immunogenicity of M701 will be assessed by summarizing the number of subjects who develop detectable anti-drug antibodies (ADAs).
Expression levels of CEA | From the time of screening period until disease progression or toxicity intolerance (up to 6 months and 14 days).
  As tumor marker, expression levels of CEA will be tested in each study site.
Expression levels of CA125 | From the time of screening period until disease progression or toxicity intolerance (up to 6 months and 14 days).
  As tumor marker, expression levels of CA125 will be tested in each study site.
Expression levels of CA72-4 | From the time of screening period until disease progression or toxicity intolerance (up to 6 months and 14 days).
  As tumor marker, expression levels of CA72-4 will be tested in each study site.
Expression levels of CA19-9 | From the time of screening period until disease progression or toxicity intolerance (up to 6 months and 14 days).
  As tumor marker, expression levels of CA19-9 will be tested in each study site.
Expression levels of AFP | From the time of screening period until disease progression or toxicity intolerance (up to 6 months and 14 days).
  As tumor marker, expression levels of AFP will be tested in each study site.
Cytokines | From the time of first dosing (Day 1) until disease progression or toxicity intolerance (up to 6 months).
  The levels of pharmacodynamic cytokines will be determined at the PD central laboratory.
Counts of Lymphocyte subsets | From the time of first dosing (Day 1) until disease progression or toxicity intolerance (up to 6 months).
  Lymphocyte subsets will be determined at the PD central laboratory.
Ascites volume | From the time of first dosing (Day 1) until disease progression or toxicity intolerance (up to 6 months).
  Ascites volume will be collected before each dose.

CONTACTS AND LOCATIONS:
Overall Officials: Jianming Xu, Principal Investigator — 307 Hospital of PLA; Shixuan Wang, Principal Investigator — Tongji Hospital
Locations (2):
- China (2):
  - The 307th Hospital of Chinese People's Liberation Army, Beijing, Beijing Municipality
  - Tongji Hospital of Tongji Medical College,Huazhong University of Science and Technology, Wuhan, Hubei

IPD SHARING:
Plan to Share IPD: No